CLINICAL TRIAL: NCT01717313
Title: A Multicenter, Phase III, Randomized, Placebo-Controlled Trial to Assess the Safety and Efficacy of MK-3102 Monotherapy in Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control
Brief Title: A Study to Assess the Safety and Efficacy of Omarigliptin (MK-3102) in Participants With Type 2 Diabetes Mellitus (T2DM) and Inadequate Glycemic Control (MK-3102-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-011; 2012-003626-24 (EudraCT Number)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin (Experimental): Omarigliptin 25 mg capsule administered orally once a week for 24 weeks (Phase A) followed by omarigliptin 25 mg administered orally once a week plus placebo to metformin daily (Phase B). Open-label metformin daily was to be initiated for participants meeting protocol-specified glycemic criteria during Phase A, but was otherwise prohibited. Open-label glimepiride daily may be initiated as glycemic rescue therapy during Phase B.
  Interventions: Drug: Omarigliptin; Drug: Metformin; Drug: Placebo to metformin; Drug: Glimepiride
- Placebo to Omarigliptin (Placebo Comparator): Placebo to omarigliptin administered orally once a week for 24 weeks (Phase A) followed by placebo to omarigliptin administered orally once a week plus metformin daily for an additional 30 weeks (Phase B). Open-label metformin was to be initiated for participants meeting protocol-specified glycemic criteria during Phase A, but was otherwise prohibited. Open-label glimepiride daily may be initiated as glycemic rescue therapy during Phase B.
  Interventions: Drug: Placebo to Omarigliptin; Drug: Metformin; Drug: Glimepiride

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin 25 mg capsule administered orally once a week.
  Arms: Omarigliptin
Drug: Placebo to Omarigliptin — Placebo to omarigliptin capsule administered orally once a week
  Arms: Placebo to Omarigliptin
Drug: Metformin — If necessary, participants may have glycemic rescue therapy initiated with open-label metformin during Phase A of the study. Participants in the placebo treatment group who were not rescued with open-label metformin during Phase A will receive blinded metformin (starting at 500 mg orally twice daily with up-titration to 1000 mg orally twice daily) in Phase B. Participants in the omarigliptin treatment group who were rescued with open-label metformin in Phase A will continue open-label metformin during Phase B of the study.
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®; Metgluco®; Glycoran®
Drug: Placebo to metformin — During Phase B of the study, participants in the omarigliptin treatment group who did not initiate glycemic rescue therapy during Phase A will receive placebo to metformin for 30 weeks (Phase B of the study).
  Arms: Omarigliptin
Drug: Glimepiride — If necessary during Phase B of the study, participants will initiate open-label glimepiride as glycemic rescue therapy
  Other Names: Armaryl®

SUMMARY:
The purpose of this study is to assess the safety and efficacy of omarigliptin (MK-3102), dosed once-weekly in participants with T2DM who have inadequate glycemic control on diet and exercise. The primary hypothesis is that after 24 weeks, treatment with omarigliptin compared with placebo provides greater reduction in hemoglobin A1c (A1C).

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Participants in India must be ≤65 years of age
* Meets one of the following criteria: currently not on an antihyperglycemic agent (AHA) for >= 12 weeks and has an A1C of >=7% and <=10% or on stable AHA monotherapy or low-dose combination therapy for > 12 weeks and has an A1C of >=6.5% and <=9%
* Participant is one of the following: male, female who is not of reproductive potential, female of reproductive potential who agrees to remain abstinent from heterosexual activity or use (or have their partner use) acceptable contraception to prevent pregnancy during the study and for 21 days after the last dose of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Has been treated with: a thiazolidinedione (TZD) within 4 months of study participation, a glucagon-like peptide-1 (GLP-1) receptor mimetic or agonist or dipeptidyl peptidase IV (DPP-4) inhibitor within 6 months of study participation, insulin or sodium-glucose cotransporter inhibitor within 12 weeks of study participation, omarigliptin at any time prior to study participation
* History of hypersensitivity to DPP-4 inhibitor
* History of intolerance, hypersensitivity or any contraindication to metformin and/or glimepiride or other sulfonylurea
* Is on a weight loss program and not in the maintenance phase or has started a weight loss medication in the past 6 months or has undergone bariatric surgery within 12 months prior to study participation
* Has undergone a surgical procedure within 4 weeks of study participation or has planned major surgery during the study
* Is on or likely to require treatment for ≥14 consecutive days or repeated courses of corticosteroids (inhaled, nasal and topical corticosteroids are permitted)
* Is currently being treated for hyperthyroidism or is on thyroid hormone therapy and has not been on a stable dose for at least 6 weeks
* Is expecting to undergo hormonal therapy in preparation to donate eggs during the study, including 21 days following the last dose of study drug
* History of active liver disease (other than non-alcoholic steatosis) including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV)
* Has had new or worsening coronary heart disease or congestive heart failure within the past 3 months, or has any of the following disorders within the past 3 months: acute coronary syndrome, coronary artery intervention, stroke or transient ischemic neurological disorder
* Has poorly controlled hypertension
* History of malignancy <=5 years prior to study participation, except for basal cell or squamous cell skin cancer or in situ cervical cancer
* Hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Pregnant or breastfeeding, or is expecting to conceive during the study, including 21 days following the last dose of study drug
* User of recreational or illicit drugs or has had a recent history of drug abuse
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking
* Has donated blood products or has had a phlebotomy within 8 weeks of study participation, or intends to donate blood products during the study or has received, or is anticipated to receive, blood products within 12 weeks of study participation or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Home P, Shankar RR, Gantz I, Iredale C, O'Neill EA, Jain L, Pong A, Suryawanshi S, Engel SS, Kaufman KD, Lai E. A randomized, double-blind trial evaluating the efficacy and safety of monotherapy with the once-weekly dipeptidyl peptidase-4 inhibitor omarigliptin in people with type 2 diabetes. Diabetes Res Clin Pract. 2018 Apr;138:253-261. doi: 10.1016/j.diabres.2017.10.018. Epub 2017 Oct 24. PMID 29079379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The double-blind treatment period included a 24-week placebo-controlled (omarigliptin/omarigliptin-matching placebo) period (Phase A) and a 30-week active-controlled period with blinded metformin/metformin matching placebo (Phase B).
Period: Phase A (Weeks 0 to 24)
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Started | 165 | 164
Completed | 147 | 151
Not Completed | 18 | 13
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Adverse Event | 4 | 2
Not completed — Non-Compliance with Study Drug | 1 | 1
Period: Interphase
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Started | 147 | 151
Completed | 146 | 151
Not Completed | 1 | 0
Not completed — Completed Phase A Did Not Enter Phase B | 1 | 0
Period: Phase B (Weeks 24 to 54)
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Started | 146 | 151
Completed | 134 | 135
Not Completed | 12 | 16
Not completed — Study Terminated by Sponsor | 4 | 4
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin | Placebo to Omarigliptin | Total
Number analyzed (Participants) | 165 | 164 | 329
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (9.2) | 57.0 (9.7) | 57.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 67 | 137
  Male | 95 | 97 | 192

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24 (Phase A, FAS Population)
Description: A1C (%) is used to report average blood glucose levels over prolonged periods of time.
  Because it was discovered that in another omarigliptin study (MK-3102-028, NCT01814748) subjects had taken metformin (prohibited per protocol, and taken without investigator knowledge), after unblinding of Phase A of this study, an analysis of metformin levels was performed on stored Week 18 blood samples. Of the subjects not rescued with metformin prior to Week 18, 10% in the omarigliptin group and 20% in the placebo group had levels showing that they were taking metformin (prohibited per protocol). The use of prohibited metformin disproportionately by the placebo group may have resulted in a smaller than expected treatment effect for efficacy outcome measures (see post-hoc analysis).
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) population was comprised of all participants who received at least one dose of study treatment and have a baseline measurement for the analysis endpoint and a post-randomization measurement for the analysis endpoint after at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percent | -0.49 [-0.73 to -0.24] | -0.10 [-0.34 to 0.14]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Terms for treatment, time, prior antihyperglycemic agent (AHA) therapy status, interaction of time by treatment, and time by prior AHA therapy status; Difference in the least squares means = -0.39, 95% CI 2-sided [-0.59 to -0.19]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event in Phase A (Excluding Data After Glycemic Rescue, Safety Population)
Description: An adverse event is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. Adverse events may include the onset of new illness and the exacerbation of preexisting conditions.
  This analysis may have been confounded by use of prohibited metformin (see results above for description of the use of prohibited metformin).
Time Frame: Up to 27 weeks
Population: The All-Participants-as-Treated (APaT) population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 41.8 | 50.0
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; Differences in percentages vs. placebo = -8.2, 95% CI 2-sided [-18.8 to 2.6]

3. Primary Outcome: Percentage of Participants Who Discontinued From the Study Drug Due to an Adverse Event in Phase A (Excluding Data After Glycemic Rescue, Safety Population)
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: The APaT population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 2.4 | 1.8
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; Difference in percentages vs. placebo = 0.6, 95% CI 2-sided [-3.1 to 4.5]

4. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (Phase A + Phase B, Excluding Data After Glycemic Rescue, Safety Population)
Description: as for outcome 2
Time Frame: Up to 57 weeks
Population: The APaT population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 54.5 | 60.4
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; Difference in percentages vs. placebo = -5.8, 95% CI 2-sided [-16.4 to 4.9]

5. Primary Outcome: Percentage of Participants Who Discontinued From the Study Drug Due to an Adverse Event (Phase A + Phase B, Excluding Data After Glycemic Rescue, Safety Population)
Description: as for outcome 2
Time Frame: Up to 57 weeks
Population: The APaT population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 3.0 | 2.4
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; Difference in percentages vs. placebo = 0.6, 95% CI 2-sided [-3.5 to 4.8]

6. Secondary Outcome: Percentage of Participants Who Achieve an A1C Goal of <7% (53 mmol/Mol) at Week 24 (Phase A, FAS Population)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). The percentage of participants who achieved A1C values <7.0% (53 mmol/mol) in the FAS population at Week 24.
  Because it was discovered that in another omarigliptin study (MK-3102-028, NCT01814748) subjects had taken metformin (prohibited per protocol, and taken without investigator knowledge), after unblinding of Phase A of this study, an analysis of metformin levels was performed on stored Week 18 blood samples. Of the subjects not rescued with metformin prior to Week 18, 10% in the omarigliptin group and 20% in the placebo group had levels showing that they were taking metformin (prohibited per protocol). The use of prohibited metformin disproportionately by the placebo group may have resulted in a smaller than expected treatment effect for efficacy outcome measures (see post-hoc analysis).
Time Frame: Week 24
Population: The FAS population was comprised of all participants who received at least one dose of study treatment and have a baseline measurement for the analysis endpoint and a post-randomization measurement for the analysis endpoint after at least one dose of study treatment, and estimated using standard multiple imputation techniques.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 36.5 [29.3 to 44.5] | 16.3 [11.3 to 22.9]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen method; Between-group rate difference = 20.3, 95% CI 2-sided [10.5 to 29.8]

7. Secondary Outcome: Percentage of Participants Who Achieve an A1C Goal of <6.5% (48 mmol/Mol) at Week 24 (Phase A, FAS Population)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). The percentage of participants who achieved A1C values <6.5% (48 mmol/mol) in the FAS population at Week 24.
  Because it was discovered that in another omarigliptin study (MK-3102-028, NCT01814748) subjects had taken metformin (prohibited per protocol, and taken without investigator knowledge), after unblinding of Phase A of this study, an analysis of metformin levels was performed on stored Week 18 blood samples. Of the subjects not rescued with metformin prior to Week 18, 10% in the omarigliptin group and 20% in the placebo group had levels showing that they were taking metformin (prohibited per protocol). The use of prohibited metformin disproportionately by the placebo group may have resulted in a smaller than expected treatment effect for efficacy outcome measures (see post-hoc analysis).
Time Frame: Week 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 16.4 [11.4 to 23.1] | 5.0 [2.5 to 9.6]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p = 0.001, Miettinen & Nurminen method; Between-group rate difference = 11.4, 95% CI 2-sided [4.8 to 18.6]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Phase A, FAS Population)
Description: Blood glucose was measured on a fasting basis (collected after an 10-hour fast). FPG is expressed as mg/dL. This change from baseline reflects the FPG level at Week 24 minus the FPG level at Week 0.
  Because it was discovered that in another omarigliptin study (MK-3102-028, NCT01814748) subjects had taken metformin (prohibited per protocol, and taken without investigator knowledge), after unblinding of Phase A of this study, an analysis of metformin levels was performed on stored Week 18 blood samples. Of the subjects not rescued with metformin prior to Week 18, 10% in the omarigliptin group and 20% in the placebo group had levels showing that they were taking metformin (prohibited per protocol). The use of prohibited metformin disproportionately by the placebo group may have resulted in a smaller than expected treatment effect for efficacy outcome measures (see post-hoc analysis).
Time Frame: Baseline and Week 24
Population: The FAS population was comprised of all participants who received at least one dose of study treatment and have a baseline measurement or a post-randomization measurement for the analysis endpoint after at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
mg/dL | -12.8 [-25.2 to -0.3] | -2.5 [-15.0 to 10.1]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p = 0.036, Constrained Longitudinal Data Analysis; Terms for treatment, time, prior AHA therapy status, the interaction of time by treatment, and time by prior AHA therapy status; Difference in the least squares means = -10.3, 95% CI 2-sided [-19.9 to -0.7]

9. Secondary Outcome: Change From Baseline in 2-hour Post Meal Glucose (PMG) at Week 24 (Phase A, FAS Population)
Description: Blood glucose was measured 2 hours after a meal (2-hour PMG). 2-hour PMG is expressed as mg/dL. This change from baseline in 2-hour PMG reflects the Week 24 2-hour PMG minus the Week 0 2-hour PMG.
  Because it was discovered that in another omarigliptin study (MK-3102-028, NCT01814748) subjects had taken metformin (prohibited per protocol, and taken without investigator knowledge), after unblinding of Phase A of this study, an analysis of metformin levels was performed on stored Week 18 blood samples. Of the subjects not rescued with metformin prior to Week 18, 10% in the omarigliptin group and 20% in the placebo group had levels showing that they were taking metformin (prohibited per protocol). The use of prohibited metformin disproportionately by the placebo group may have resulted in a smaller than expected treatment effect for efficacy outcome measures (see post-hoc analysis).
Time Frame: Baseline and Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 106 | 102
mg/dL | -25.6 [-56.0 to 4.8] | -13.9 [-43.5 to 15.6]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p = 0.177, Constrained Longitudinal Data Analysis; [statistical method as in outcome 8, analysis 1]; Difference in the least squares means = -11.6, 95% CI 2-sided [-28.6 to 5.3]

10. Secondary Outcome: Change From Baseline in A1C at Week 54 (Phase A + Phase B, FAS Population)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Thus, this change from baseline reflects the Week 54 A1C minus the Week 0 A1C.
  The results of the study at Week 54 may have been confounded by use of prohibited metformin (see results above for description of the use of prohibited metformin).
Time Frame: Baseline and Week 54
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percent | -0.40 [-0.67 to -0.13] | -0.80 [-1.07 to -0.53]

11. Secondary Outcome: Percentage of Participants Who Achieve an A1C Goal of <7% (53 mmol/Mol) at Week 54 (Phase A + Phase B, FAS Population)
Description: The percentage of participants who achieved A1C values <7.0% (53 mmol/mol) in the FAS population at Week 54.
  The results of the study at Week 54 may have been confounded by use of prohibited metformin (see results above for description of the use of prohibited metformin).
Time Frame: Week 54
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 33.8 [26.8 to 41.5] | 43.8 [36.2 to 51.7]

12. Secondary Outcome: Percentage of Participants Who Achieve an A1C Goal of <6.5% at Week 54 (Phase A + Phase B, FAS Population)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). The percentage of participants who achieved A1C values <6.5% (48 mmol/mol) in the FAS population at Week 54.
  The results of the study at Week 54 may have been confounded by use of prohibited metformin (see results above for description of the use of prohibited metformin).
Time Frame: Week 54
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
Percentage of participants | 14.5 [9.7 to 21.2] | 20.6 [14.8 to 28.0]

13. Secondary Outcome: Change From Baseline in FPG at Week 54 (Phase A + Phase B, FAS Population)
Description: Blood glucose was measured on a fasting basis (collected after an 10-hour fast). FPG is expressed as mg/dL. This change from baseline reflects the FPG level at Week 54 minus the FPG level at Week 0.
  The results of the study at Week 54 may have been confounded by use of prohibited metformin (see results above for description of the use of prohibited metformin).
Time Frame: Baseline and Week 54
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 165 | 164
mg/dL | -8.3 [-19.8 to 3.2] | -21.1 [-32.7 to -9.5]

14. Post Hoc Outcome: Change From Baseline in A1C at Week 24 (Phase A, Per-Protocol Population)
Description: A1C is a blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Thus, this change from baseline reflects the Week 24 A1C minus the Week 0 A1C.
  A post-hoc sensitivity analysis was performed that excluded participants in both treatment groups who were found to have used prohibited metformin (see results above for a description of the use of prohibited metformin).
Time Frame: Baseline and Week 24
Population: The Per-Protocol population excluded participants from the FAS population who either had <75% drug compliance or used a prohibited medication (including metformin).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 149 | 131
Percent | -0.54 [-0.68 to -0.39] | -0.00 [-0.17 to 0.16]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 8, analysis 1]; Difference in the least squares means = -0.53, 95% CI 2-sided [-0.75 to -0.32]

15. Post Hoc Outcome: Change From Baseline in FPG at Week 24 (Phase A, Per-Protocol Population)
Description: Blood glucose was measured on a fasting basis (collected after an 10-hour fast). FPG is expressed as mg/dL. This change from baseline reflects the FPG level at Week 24 minus the FPG level at Week 0.
  A post-hoc sensitivity analysis was performed that excluded participants in both treatment groups who were found to have used prohibited metformin (see results above for a description of the use of prohibited metformin).
Time Frame: Baseline and Week 24
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 149 | 131
mg/dL | -15.5 [-22.5 to -8.4] | -2.2 [-10.9 to 6.4]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p = 0.014, Constrained Longitudinal Data Analysis; [statistical method as in outcome 8, analysis 1]; Difference in the least squares means = -13.2, 95% CI 2-sided [-23.7 to -2.7]

16. Post Hoc Outcome: Change From Baseline in 2-hour PMG at Week 24 (Phase A, Per-Protocol Population)
Description: Blood glucose was measured 2 hours after a meal (2-hour PMG). 2-hour PMG is expressed as mg/dL. This change from baseline in 2-hour PMG reflects the Week 24 2-hour PMG minus the Week 0 2-hour PMG.
  A post-hoc sensitivity analysis was performed that excluded participants in both treatment groups who were found to have used prohibited metformin (see results above for a description of the use of prohibited metformin).
Time Frame: Baseline and Week 24
Population: The Per Protocol population excluded participants from the FAS population who either had <75% drug compliance or used a prohibited medication (including metformin).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Number analyzed (Participants) | 95 | 80
mg/dL | -40.1 [-53.4 to -26.9] | -19.6 [-34.1 to -5.2]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo to Omarigliptin; Test type: Superiority or Other; p = 0.031, Constrained Longitudinal Data Analysis; [statistical method as in outcome 8, analysis 1]; Difference in the least squares means = -20.5, 95% CI 2-sided [-39.0 to -1.9]

ADVERSE EVENTS:
Time Frame: Up to 57 weeks for serious adverse events (SAE, including 3-week follow-up) and up to 54 weeks for non-serious adverse events.
Description: SAE tables include data after glycemic rescue. Non-SAE tables exclude data after glycemic rescue.
  This analysis may have been confounded by use of prohibited metformin (see use of prohibited metformin).
Arm/Group | Omarigliptin | Placebo to Omarigliptin
Serious Adverse Events (participants affected / at risk) | 8/165 | 8/164
Other Adverse Events (participants affected / at risk) | 31/165 | 25/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=165) | Placebo to Omarigliptin (N=164)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=165) | Placebo to Omarigliptin (N=164)
Nasopharyngitis (Infections and infestations) | 17 (21) | 12 (16)
Blood glucose increased (Investigations) | 14 (14) | 13 (13)

LIMITATIONS AND CAVEATS:
Care must be taken in the interpretation of the results in this study as the non-protocol-specified prohibited use of metformin among a number of participants may have impacted the safety and efficacy results disproportionally among study arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.